CLINICAL TRIAL: NCT03856112
Title: A Phase 1/2 Study of MLN9708 (Ixazomib [I]), Venetoclax (V), and Dexamethasone (D) Regimen (IVD) to Restore or Enhance Proteasome Inhibitor (PI) Sensitivity in Non-t(11;14) Relapsed/Refractory Multiple Myeloma (RRMM)
Brief Title: Ixazomib and Dexamethasone With or Without Venetoclax in Treating Patients With Non-t(11;14) Relapsed or Refractory Multiple Myeloma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Per CTEP, Martha Khrum this study is withdrawn. Changing status to update CT.gov
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-00994; NCI-2019-00994 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10248 (Other: University Health Network Princess Margaret Cancer Center LAO); 10248 (Other: CTEP); UM1CA186644 (NIH)
Record Dates: First submitted 2019-02-22; First posted 2019-02-27 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma; t(11;14) Negative
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; ixazomib; MLN2238; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (ixazomib, venetoclax, dexamethasone) (Experimental): Patients receive ixazomib citrate PO on days 1, 8, and 15, venetoclax PO QD on days 1-28 and dexamethasone PO on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Drug: Ixazomib; Drug: Ixazomib Citrate; Drug: Venetoclax
- Arm II (ixazomib, dexamethasone) (Active Comparator): Patients receive ixazomib citrate PO on days 1, 8, and 15, and dexamethasone PO on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Drug: Ixazomib; Drug: Ixazomib Citrate
- Arm III (ixazomib, venetoclax, dexamethasone) (Experimental): PI-refractory patients receive ixazomib citrate, venetoclax and dexamethasone as Arm I.
  Interventions: Drug: Dexamethasone; Drug: Ixazomib; Drug: Ixazomib Citrate; Drug: Venetoclax

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Ixazomib — Given PO
  Other Names: MLN-2238; MLN2238
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN-9708; MLN9708; Ninlaro
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta
  Arms: Arm I (ixazomib, venetoclax, dexamethasone); Arm III (ixazomib, venetoclax, dexamethasone)

SUMMARY:
This phase I/II trial studies the best dose and side effects of venetoclax and how well it works in combination with ixazomib and dexamethasone in treating patients with t(11;14) negative multiple myeloma that has come back or does not respond to treatment. Ixazomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as venetoclax and dexamethasone work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known how well venetoclax works with ixazomib and dexamethasone in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety profile and tolerability of oral combination therapy with ixazomib citrate (ixazomib) (I), venetoclax (V), dexamethasone (D) in non-t(11;14) relapsed/refractory multiple myeloma (RRMM) with dose-escalating design to determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D). (Phase I) II. To compare overall response rate (ORR; measured as best response) of IVD and ID in a proteasome inhibitor (PI)-non-refractory cohort. (Phase II, Cohort 1) III. To evaluate ORR of IVD in PI-refractory cohort. (Phase II, Cohort 2)

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To determine the rate of very good partial response (VGPR) or better. III. To determine time to progression (TTP). IV. To determine duration of response (DOR). V. To determine progression-free survival (PFS). VI. To determine overall survival (OS).

EXPLORATORY OBJECTIVES:

I. To correlate and predict responses with the following tests, using bone marrow aspirate samples at (a) baseline and (b) during treatment on day 8 (or day 9 to allow for scheduling flexibility): BCL2, NOXA, and MCL1 by flow cytometry; polymerase chain reaction (PCR) for BCL2, BCL2L1 (=BCL-XL), and MCL-1 messenger ribonucleic acid (mRNA) expression, and BCL2:BCL2L1 and BCL2:MCL1 ratios; and Ex vivo Mathematical Myeloma Advisor (EMMA).

II. To evaluate the drug exposure and to correlate with toxicities using venetoclax peripheral blood pharmacokinetic (PK) analysis.

OUTLINE: This is a phase I, dose-escalation study of venetoclax followed by a phase II study. PI non-refractory patients are randomized to 1 of 2 arms.

ARM I: Patients receive ixazomib citrate orally (PO) on days 1, 8, and 15, venetoclax PO once daily (QD) on days 1-28 and dexamethasone PO on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive ixazomib citrate PO on days 1, 8, and 15, and dexamethasone PO on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM III: PI-refractory patients receive ixazomib citrate, venetoclax and dexamethasone as Arm I.

After completion of study treatment, patients are followed for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* ELIGIBILITY CRITERIA FOR PHASE I AND PHASE II
* Patients must have RRMM without t(11;14), confirmed by fluorescence in situ hybridization (FISH).
* RRMM with measurable disease with at least one of the following: M-protein >= 0.5 g/dL in serum or >= 200 mg/24-hour in urine, or serum free light chain (FLC) >= 10 mg/dL with abnormal serum FLC ratio for subjects without measurable disease by serum protein electrophoresis (SPEP) or urine protein electrophoresis (UPEP) criteria.
* Prior multiple myeloma (MM) treatment:

  * Received at least 2 lines of prior therapy (including at least one PI, excluding MLN9708), or
  * Received 1 prior line of therapy with both a PI (excluding MLN9708) and an immunomodulatory (IMiD) agent.
* PI-refractory (only applicable to phase 2, cohort 2): progressing =< 60 days of the last PI therapy or < 25% response while on therapy.
* PI-non-refractory (only applicable to phase 2, cohort 1): not meeting PI-refractory criteria, i.e., (a) did not progress =< 60 days of the last PI therapy and (b) had >= 25% response while on therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%).
* Absolute neutrophil count (ANC) >= 1,000/mcL (patients may not use growth factor support to achieve ANC criteria for eligibility assessment).
* Platelets >= 50,000/mcL (patients may not receive a platelet transfusion within 72 hours of eligibility assessment).
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN).
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional ULN.
* Calculated creatinine clearance >= 30 mL/min (measured by either 24-hour urine collection or calculated using the Cockcroft-Gault formula).
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have completed treatment previously and cured (i.e., undetectable HCV viral load).
* Patients with treated brain metastases are eligible if there is no evidence of progression for at least 4 weeks after central nervous system (CNS)- directed treatment, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT] scan) during the screening period.
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate central nervous system (CNS) specific treatment is not required and is unlikely to be required for at least 4 weeks (or scheduled assessment after the first cycle of treatment), and a risk-benefit analysis (discussion) by the patient and the investigator favors participation in the clinical trial.
* The effects of MLN9708 and venetoclax in combination with dexamethasone on the developing human fetus are unknown. For this reason and because corticosteroids like dexamethasone are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 3 months after completion of the administration of the study agents. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.
* Known human immunodeficiency virus (HIV)-positive patients who meet the following criteria will be considered eligible:

  * CD4 count > 350 cells/mm^3
  * Undetectable viral load
  * Maintained on modern therapeutic regimens (utilizing non-CYP-interactive agents)
  * No history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections.

Exclusion Criteria:

* Patients who have been previously treated with MLN9708 or venetoclax or other direct BCL2 inhibitor.
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities grade > 1), except for grade 2 peripheral sensory neuropathy.
* Patients who are receiving any other anti-myeloma chemotherapy or radiotherapy, immunotherapy, or investigational agents within 2 weeks or 5 half-lives (whichever is longer and/or applicable) of the start of the trial.
* Patients receiving dexamethasone >= 40 mg/day or equivalent of any corticosteroids within 2 weeks of the start of the trial.
* Patients with non-secretory MM, plasma cell leukemia (i.e., >= 20% plasma cells in peripheral blood differential or >= 2,000/mcL circulating plasma cells), symptomatic primary light chain (AL) amyloidosis, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
* Prior allogeneic hematopoietic cell transplantation (HCT) within the last 12 months and evidence of active graft-versus-host disease (GVHD).
* Prior autologous HCT within the last 3 months.
* History of active malignancies other than MM within the last 2 years unless treated with curative intent and has no evidence of active disease. Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin are excluded from this criterion.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MLN9708, venetoclax, or dexamethasone. This includes boron and boron-containing products.
* Patients requiring chronic administration of any medications or substances that are strong inhibitors or inducers of CYP3A4 enzyme are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* Patients with uncontrolled intercurrent illness.
* Female patients who are lactating or have a positive serum pregnancy test during the screening period are excluded from this study because MLN9708 is a proteasome inhibitor with the potential for embryo-lethal effects, and an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with MLN9708. Patients must stop breastfeeding while on MLN9708 and until 90 days have passed since their last dose. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-21 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose/recommended phase II dose (MTD/RP2D) of venetoclax (Phase I) | Up to 28 days
  The MTD is defined as the highest dose level in which 1 or fewer of 6 patients experience a dose limiting toxicity. That dose level is considered the MTD/RP2D.
Overall response rate (ORR) (Phase II) | Up to 2.5 years
  For cohort 1, the difference in ORR between the two arms will be tested by using the Cochran-Mantel-Haenszel (CMH) test.
Overall response rate (ORR) (Phase II) | Up to 2.5 years
  For cohort 2, the ORR will be estimated, and the lower limit of the one-sided 90% confidence interval (CI) will be computed using the Atkinson and Brown method (Atkinson and Brown 1985), which accounts for the nature of a two-stage design.

SECONDARY OUTCOMES:
Very good partial response (VGPR) or better response rate | Up to 2.5 years
  VGPR or better response rate is defined as the proportion of subjects with documented VGPR or better based on the International Myeloma Working Group criteria. The binomial distribution will be used to calculate the point estimate of the VGPR or better response rate and 95% CI for each study arm. The difference in VGPR or better response rate between two arms in cohort 1 will be assessed by the CMH test.
Time to progression (TTP) | From the date of the first dose of study drug (cohort 2) or date of randomization (cohort 1) to the date of first documented progressive disease (PD) or death due to multiple myeloma, whichever occurs first, assessed up to 2.5 years
  Kaplan-Meier plots will be presented for TTP.
Time to progression (TTP) | From the date of the first dose of study drug (cohort 2) or date of randomization (cohort 1) to the date of first documented PD or death due to multiple myeloma, whichever occurs first, assessed up to 2.5 years
  The difference between ixazomib, venetoclax, dexamethasone (IVD) and ixazomib, dexamethasone (ID) in cohort 1 will be assessed by the stratified log-rank test.
Time to progression (TTP) | From the date of the first dose of study drug (cohort 2) or date of randomization (cohort 1) to the date of first documented PD or death due to multiple myeloma, whichever occurs first, assessed up to 2.5 years
  The hazard ratio of time-to-event endpoints for IVD versus ID in cohort 1 will be estimated by the stratified Cox proportional hazard regression model.
Progression-free survival (PFS) | From the date of the first dose of study drug (cohort 2) or date of randomization (cohort 1) to the date of first documented PD or death due to any cause, whichever occurs first, assessed up to 2.5 years
  Kaplan-Meier plots will be presented for PFS.
Progression-free survival (PFS) | From the date of the first dose of study drug (cohort 2) or date of randomization (cohort 1) to the date of first documented PD or death due to any cause, whichever occurs first, assessed up to 2.5 years
  The difference between IVD and ID in cohort 1 will be assessed by the stratified log-rank test.
Progression-free survival (PFS) | From the date of the first dose of study drug (cohort 2) or date of randomization (cohort 1) to the date of first documented PD or death due to any cause, whichever occurs first, assessed up to 2.5 years
  The hazard ratio of time-to-event endpoints for IVD versus ID in cohort 1 will be estimated by the stratified Cox proportional hazard regression model.
Duration of response (DOR) | From the subject's date of first documented response (partial response [PR] or better) to the date of first documented PD or death due to multiple myeloma (MM), whichever occurs first, assessed up to 2.5 years
  Kaplan-Meier plots will be presented for DOR.
Duration of response (DOR) | From the subject's date of first documented response (PR or better) to the date of first documented PD or death due to MM, whichever occurs first, assessed up to 2.5 years
  The difference between IVD and ID in cohort 1 will be assessed by the stratified log-rank test.
Duration of response (DOR) | From the subject's date of first documented response (PR or better) to the date of first documented PD or death due to MM, whichever occurs first, assessed up to 2.5 years
  The hazard ratio of time-to-event endpoints for IVD versus ID in cohort 1 will be estimated by the stratified Cox proportional hazard regression model.
Overall survival (OS) | From the subject's date of the first dose of study drug (cohort 2) or date of randomization (cohort 1) to the date of death due to any cause, assessed up to 2.5 years
  Kaplan-Meier plots will be presented for OS.
Overall survival (OS) | From the subject's date of the first dose of study drug (cohort 2) or date of randomization (cohort 1) to the date of death due to any cause, assessed up to 2.5 years
  The difference between IVD and ID in cohort 1 will be assessed by the stratified log-rank test.
Overall survival (OS) | From the subject's date of the first dose of study drug (cohort 2) or date of randomization (cohort 1) to the date of death due to any cause, assessed up to 2.5 years
  The hazard ratio of time-to-event endpoints for IVD versus ID in cohort 1 will be estimated by the stratified Cox proportional hazard regression model.

OTHER OUTCOMES:
BCL2 biomarker analysis | At screening and day 8
  The association between ORR and the change from screening to day 8 will be assessed by the Satterthwaite t-test if the normality assumption is met.
BCL2 biomarker analysis | At screening and day 8
  The association with baseline measures will be explored. The data transformation may be employed to use the parametric analytic tools. If the assumption is not met, the non-parametric alternatives such as the Wilcoxon rank-sum test will be used. No multiplicity adjustment is planned for exploratory biomarkers analysis.
NOXA biomarker analysis | At screening and day 8
  The association between ORR and the change from screening to day 8 will be assessed by the Satterthwaite t-test if the normality assumption is met.
NOXA biomarker analysis | At screening and day 8
  The association with baseline measures will be explored. The data transformation may be employed to use the parametric analytic tools. If the assumption is not met, the non-parametric alternatives such as the Wilcoxon rank-sum test will be used. No multiplicity adjustment is planned for exploratory biomarkers analysis.
MCL1 biomarker analysis | At screening and day 8
  The association between ORR and the change from screening to day 8 will be assessed by the Satterthwaite t-test if the normality assumption is met.
MCL1 biomarker analysis | At screening and day 8
  The association with baseline measures will be explored. The data transformation may be employed to use the parametric analytic tools. If the assumption is not met, the non-parametric alternatives such as the Wilcoxon rank-sum test will be used. No multiplicity adjustment is planned for exploratory biomarkers analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Taiga Nishihori, Principal Investigator — University Health Network Princess Margaret Cancer Center LAO